CLINICAL TRIAL: NCT06302426
Title: An Open-label, Multiple-Ascending Dose, Two-Part Dose Ranging and Cohort Expansion Study of INI-4001 in Patients With Advanced Solid Tumours
Brief Title: Trial of INI-4001 in Patients With Advanced Solid Tumours
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Inimmune Corporation (Industry)
Collaborators: Avance Clinical Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INI-4001-101
Record Dates: First submitted 2024-01-16; First posted 2024-03-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Nivolumab; pembrolizumab; cemiplimab; avelumab; atezolizumab; durvalumab

STUDY DESIGN:
Intervention Model Description: This is a Phase Ia/Ib, open-label, dose-escalation and dose expansion study. This study will be conducted in two parts: Phase Ia (dose escalation) and Phase Ib (dose expansion).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- INI-4001 Monotherapy Dose Escalation - INI-4001 Dose Level 1 (Experimental): For dose-level 1, INI-4001 will be administered intravenously once per week on Days 1, 8 and 15 of a 21-day cycle. A complementary therapy may be introduced in combination with INI-4001.
  Interventions: Drug: INI-4001; Combination Product: Nivolumab; Combination Product: Pembrolizumab; Combination Product: Cemiplimab; Combination Product: Avelumab; Combination Product: Atezolizumab; Combination Product: Durvalumab
- INI-4001 Monotherapy Dose Escalation - INI-4001 Dose Level 2 (Experimental): For dose-level 2, INI-4001 will be administered intravenously once per week on Days 1, 8 and 15 of a 21-day cycle. A complementary therapy may be introduced in combination with INI-4001.
  Interventions: Drug: INI-4001; Combination Product: Nivolumab; Combination Product: Pembrolizumab; Combination Product: Cemiplimab; Combination Product: Avelumab; Combination Product: Atezolizumab; Combination Product: Durvalumab
- INI-4001 Monotherapy Dose Escalation - INI-4001 Dose Level 3 (Experimental): For dose-level 3, INI-4001 will be administered intravenously once per week on Days 1, 8 and 15 of a 21-day cycle. A complementary therapy may be introduced in combination with INI-4001.
  Interventions: Drug: INI-4001; Combination Product: Nivolumab; Combination Product: Pembrolizumab; Combination Product: Cemiplimab; Combination Product: Avelumab; Combination Product: Atezolizumab; Combination Product: Durvalumab
- INI-4001 Monotherapy Dose Escalation - INI-4001 Dose Level 4 (Experimental): For dose-level 4, INI-4001 will be administered intravenously once per week on Days 1, 8 and 15 of a 21-day cycle. A complementary therapy may be introduced in combination with INI-4001.
  Interventions: Drug: INI-4001; Combination Product: Nivolumab; Combination Product: Pembrolizumab; Combination Product: Cemiplimab; Combination Product: Avelumab; Combination Product: Atezolizumab; Combination Product: Durvalumab
- INI-4001 Monotherapy Dose Escalation - INI-4001 Dose Level 5 (Experimental): For dose-level 5, INI-4001 will be administered intravenously once per week on Days 1, 8 and 15 of a 21-day cycle. A complementary therapy may be introduced in combination with INI-4001.
  Interventions: Drug: INI-4001; Combination Product: Nivolumab; Combination Product: Pembrolizumab; Combination Product: Cemiplimab; Combination Product: Avelumab; Combination Product: Atezolizumab; Combination Product: Durvalumab
- INI-4001 Monotherapy Dose Escalation - INI-4001 Dose Level 6 (Experimental): For dose-level 6, INI-4001 will be administered intravenously once per week on Days 1, 8 and 15 of a 21-day cycle. A complementary therapy may be introduced in combination with INI-4001.
  Interventions: Drug: INI-4001; Combination Product: Nivolumab; Combination Product: Pembrolizumab; Combination Product: Cemiplimab; Combination Product: Avelumab; Combination Product: Atezolizumab; Combination Product: Durvalumab

INTERVENTIONS:
Drug: INI-4001 — INI-4001 is a small molecule TLR7/8 agonist being developed as a standalone treatment for the induction of anti-tumour immune responses and sensitization to immune checkpoint inhibitor (ICI) therapy.
Combination Product: Nivolumab — During both Phase Ia and Phase Ib, patients may meeting required criteria (at the discretion of the PI in consultation with the study Sponsor) may transition to combination therapy.
  Other Names: Opdivo
Combination Product: Pembrolizumab — During both Phase Ia and Phase Ib, patients meeting required criteria (at the discretion of the PI in consultation with the study Sponsor) transition to combination therapy.
  Other Names: Keytruda
Combination Product: Cemiplimab — During both Phase Ia and Phase Ib, patients meeting required criteria (at the discretion of the PI in consultation with the study Sponsor) transition to combination therapy.
  Other Names: Libtayo
Combination Product: Avelumab — During both Phase Ia and Phase Ib, patients meeting required criteria (at the discretion of the PI in consultation with the study Sponsor) transition to combination therapy.
  Other Names: Bavencio
Combination Product: Atezolizumab — During both Phase Ia and Phase Ib, patients meeting required criteria (at the discretion of the PI in consultation with the study Sponsor) transition to combination therapy.
  Other Names: Tecentriq
Combination Product: Durvalumab — During both Phase Ia and Phase Ib, patients meeting required criteria (at the discretion of the PI in consultation with the study Sponsor) transition to combination therapy.
  Other Names: Imfinzi

SUMMARY:
Phase 1 open-label, dose-escalation and dose-expansion study of INI-4001 as a single agent and in combination with approved checkpoint inhibitors in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
This is a Phase Ia/Ib, open-label, dose-escalation, and dose expansion study. This study will be conducted in two parts: Phase Ia (dose escalation) and Phase Ib (dose expansion). Phase Ia will initially seek to establish the MTD of INI-4001 administered as a monotherapy. Following identification of the MTD, any dose level at or below the MTD may be further expanded to further explore the safety, PK, PD, and preliminary efficacy of INI-4001 alone and in combination with a complementary therapy (Phase Ib).

Following cessation of INI-4001, patients will be requested to participate in long-term follow-up to assess overall survival. This long-term follow-up will continue for each patient until at least 1 year after their last dose of INI-4001, or until otherwise advised by the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has locally advanced or metastatic cancer (all solid tumours allowed except primary brain/CNS tumour or untreated spinal cord compression)
2. Patient has at least one extracranial measurable disease lesion per RECIST 1.1/ iRECIST criteria.
3. Patients with known brain metastases are eligible if they meet all the following criteria:

   1. Patient has received definitive treatment of brain metastases with stereotactic body radiation therapy (SBRT) or surgery provided that the brain lesions are stable (without evidence of progression by imaging for at least 4 weeks before the first dose of study treatment)
   2. Patient is neurologically stable and has had no persistent side effects / complications from prior treatment.
   3. Patient has no evidence of new or enlarging brain metastases (confirmed by repeat imaging) and has not required steroids for at least 14 days prior to first dose administration on Day 1.
4. Female patients must be of non-child-bearing potential i.e., surgically sterilised at least 6 weeks before the screening visit or postmenopausal

Exclusion Criteria:

1. Prior therapy with a TLR7 and/or TLR8 agonist, unless first approved by the medical monitor.
2. Has primary brain/CNS tumour or untreated spinal cord compression.
3. Has known active, uncontrolled brain or CNS metastases and/or carcinomatous meningitis.
4. Evidence of abnormal cardiac function
5. Clinically significant active infection within 2 weeks prior to commencement of treatment, or unexplained fever (temperature > 38.1°C) within 7 days prior to first dose administration on Cycle 1 Day 1.
6. Known active human immunodeficiency virus (HIV-1 or HIV-2), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibodies at the screening visit.
7. History of other malignancy not meeting inclusion criterion #1 within the past 2 years
8. Major surgery within 28 days of Cycle 1, Day 1, or minor surgical procedures within 7 days of Cycle 1, Day 1.
9. Received cancer-directed therapy
10. A history of autoimmune diseases that has caused terminal organ damage or required systemic immunosuppression / systemic disease modulating drugs within the past 2 years.
11. Chronic use of immune-suppressive drugs (i.e., systemic corticosteroids used in the management of cancer or non-cancer related illnesses, (e.g., COPD) in dosing exceeding 10 mg daily of prednisone equivalent). Inhaled steroids are allowed.
12. History of prior organ allograft.
13. Known hypersensitivity to the study drug or its inactive ingredients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) during Cycle 1 to determine the maximum tolerated dose of INI-4001 Monotherapy | Assessed from Cycle 1 Day 1 through to Cycle 1 Day 21
  Graded using a 5 point scale

SECONDARY OUTCOMES:
Incidence, type, and severity of treatment-emergent adverse events (TEAEs) leading to discontinuation of study treatment after multiple ascending doses | Assessed at Screening, then daily from Cycle 1 Day 1 through to 30 days post last dose of INI-4001
  Graded using a 5 point scale
Incidence and nature of dose-limiting toxicities (DLTs) and regimen-limiting toxicities (RLTs) leading to discontinuation of study treatment after multiple ascending doses | Assessed from Cycle 1 Day 1 through to Cycle 1 Day 21
  Graded using a 5 point scale
Number of Participants with a Change from baseline in Vital signs measurements after multiple ascending doses | Assessed at Screening, then Cycle 1 Day 1 through to 30 days post last dose of INI-4001
  Pulse rate [PR], systolic and diastolic blood pressure [BP], temperature, respiratory rate.[RR] and oxygen saturation.
  Blood pressure will be measured using a sphygmomanometer, body temperature will be measured using a thermometer, Heart rate (HR) is measured using vital sign machine,respiratory rate is measured manually via 60- second count.[RR] and oxygen saturation is measured using a Oximeter. All abnormal assessments measured as Clinically significant post dose will be recorded as AEs.
Number of Participants with a Change from baseline in body weight after multiple ascending doses | Assessed at Screening then pre-dose on Day 1 of each 21 day cycle, assessed for up to 36 months or until disease progression, which occurs first
  Weight will be measured utilising scales
Number of Participants with a Change from baseline in clinical laboratory parameters (haematology) after multiple ascending doses | Assessed at Screening, then Day 1 and Day 15 of each 21 day cycle, assessed for up to 36 months or until disease progression, which occurs first
  Haematology - blood samples will be collected. All safety laboratory assessments will be assessed by a local laboratory according to their reference ranges.
Number of Participants with a Change from baseline in clinical laboratory parameters (serum chemistry) after multiple ascending doses | Assessed at Screening, then Day 1 and Day 15 of each 21 day cycle, assessed for up to 36 months or until disease progression, which occurs first
  Serum Chemistry - blood samples will be collected. All safety laboratory assessments will be assessed by a local laboratory according to their reference ranges.
Number of Participants with a Change from baseline in clinical laboratory parameters (urinalysis) after multiple ascending doses | Assessed at Screening, then Day 1 and Day 15 of each 21 day cycle, assessed for up to 36 months or until disease progression, which occurs first
  Urinalysis - urine samples will be collected. All safety laboratory assessments will be assessed by a local laboratory according to their reference ranges.
Change from baseline in measurements of HR in beats per minute after multiple ascending doses | Assessed at Screening, then Cycle 1 Day 1 through to Day 16 and then at 7 days and 30 days post last dose of INI-4001
  12-lead ECG parameters include the measurements of HR in beats per minute. 12-lead ECG will be taken in triplicate at screening and prior to infusion and as single measurements at all other timepoints.
Change from baseline in measurements of PR interval via 12-lead electrocardiogram after multiple ascending doses | Assessed at Screening, then Cycle 1 Day 1 through to Day 16 and then at 7 days and 30 days post last dose of INI-4001
  12-lead ECG parameters include the measurements of PR interval. 12-lead ECG will be taken in triplicate at screening and prior to infusion and as single measurements at all other timepoints.
Change from baseline in measurements of QT interval via 12-lead electrocardiogram after multiple ascending doses | Assessed at Screening, then Cycle 1 Day 1 through to Day 16 and then at 7 days and 30 days post last dose of INI-4001
  12-lead ECG parameters include the . 12-lead ECG will be taken in triplicate at screening and prior to infusion and as single measurements at all other timepoints.
Change from baseline in measurements of RR interval in breaths per minute via 12-lead electrocardiogram after multiple ascending doses | Assessed at Screening, then Cycle 1 Day 1 through to Day 16 and then at 7 days and 30 days post last dose of INI-4001
  12-lead ECG parameters include the measurements of RR interval in breaths per minute. 12-lead ECG will be taken in triplicate at screening and prior to infusion and as single measurements at all other timepoints.
Change from baseline in measurements of QRS duration via 12-lead electrocardiogram after multiple ascending doses | Assessed at Screening, then Cycle 1 Day 1 through to Day 16 and then at 7 days and 30 days post last dose of INI-4001
  12-lead ECG parameters include the measurements of QRS duration. 12-lead ECG will be taken in triplicate at screening and prior to infusion and as single measurements at all other timepoints.
Change from baseline in measurements of QTcF via 12-lead electrocardiogram after multiple ascending doses | Assessed at Screening, then Cycle 1 Day 1 through to Day 16 and then at 7 days and 30 days post last dose of INI-4001
  12-lead ECG parameters include the measurements of QTcF. 12-lead ECG will be taken in triplicate at screening and prior to infusion and as single measurements at all other timepoints.
Change from baseline in Eastern Cooperative Oncology Group (ECOG) score after multiple ascending doses | Screening, then Cycle 1 & Cycle 2 (each cycle is 21 days) on Day 1, Day 8 and Day 15 and then at 7 days and 30 days post last dose of INI-4001
  Graded using a 6 point scale
Single dose PK Parameters - maximum observed concentration (Cmax) | Cycle 1 Day 1 & Day 15, pre-dose, EOI (within 2 minutes), then 15 & 30 minutes, 1, 2, 4 & 6 hours post-dose, Day 2 & Day 16 at 24 hours post-dose, Cycle 2 & 4 Day 1 pre-dose, EOI, Day 8 pre-dose then 7 days post last infusion (a cycle is 21 days)
  Pharmacokinetics (PK) of INI-4001 in blood plasma following a single dose
Multiple dose PK Parameters - maximum observed concentration (Cmax) | Cycle 1 Day 1 & Day 15, pre-dose, EOI (within 2 minutes), then 15 & 30 minutes, 1, 2, 4 & 6 hours post-dose, Day 2 & Day 16 at 24 hours post-dose, Cycle 2 & 4 Day 1 pre-dose, EOI, Day 8 pre-dose then 7 days post last infusion (a cycle is 21 days)
  Pharmacokinetics (PK) of INI-4001 in blood plasma following multiple doses
Single dose PK Parameters - Time to Cmax (Tmax) | Cycle 1 Day 1 & Day 15, pre-dose, EOI (within 2 minutes), then 15 & 30 minutes, 1, 2, 4 & 6 hours post-dose, Day 2 & Day 16 at 24 hours post-dose, Cycle 2 & 4 Day 1 pre-dose, EOI, Day 8 pre-dose then 7 days post last infusion (a cycle is 21 days)
  Pharmacokinetics (PK) of INI-4001 in blood plasma following a single dose
Multiple dose PK Parameters - Time to Cmax (Tmax) | Cycle 1 Day 1 & Day 15, pre-dose, EOI (within 2 minutes), then 15 & 30 minutes, 1, 2, 4 & 6 hours post-dose, Day 2 & Day 16 at 24 hours post-dose, Cycle 2 & 4 Day 1 pre-dose, EOI, Day 8 pre-dose then 7 days post last infusion (a cycle is 21 days)
  Pharmacokinetics (PK) of INI-4001 in blood plasma following multiple doses
Single dose PK Parameters - Area under the concentration-time curve from time 0 to 24 hours post-dose (AUC0-24) | Cycle 1 Day 1 & Day 15, pre-dose, EOI (within 2 minutes), then 15 & 30 minutes, 1, 2, 4 & 6 hours post-dose, Day 2 & Day 16 at 24 hours post-dose, Cycle 2 & 4 Day 1 pre-dose, EOI, Day 8 pre-dose then 7 days post last infusion (a cycle is 21 days)
  Pharmacokinetics (PK) of INI-4001 in blood plasma following a single dose
Single dose PK Parameters - Total amount excreted in urine (Ae) | Cycle 1 Day 1 pre-dose, then 0-2, 2-4 and 4-6 hours post-dose, Day 1 to Day 2 6-24 hours post-dose (each cycle is 21 days)
  Pharmacokinetics (PK) of INI-4001 in urine following a single dose
Single dose PK Parameters - Fraction excreted in the urine (Fe) | Cycle 1 Day 1 pre-dose, then 0-2, 2-4 and 4-6 hours post-dose, Day 1 to Day 2 6-24 hours post-dose (each cycle is 21 days)
  Pharmacokinetics (PK) of INI-4001 in urine following a single dose
Single dose PK Parameters - Renal clearance (CLr) | Cycle 1 Day 1 pre-dose, then 0-2, 2-4 and 4-6 hours post-dose, Day 1 to Day 2 6-24 hours post-dose (each cycle is 21 days)
  Pharmacokinetics (PK) of INI-4001 in urine following a single dose
Multiple dose PK Parameters - Area under the concentration-time curve from time 0 to 24 hours post-dose (AUC0-24) | Cycle 1 Day 1 & Day 15, pre-dose, EOI (within 2 minutes), then 15 & 30 minutes, 1, 2, 4 & 6 hours post-dose, Day 2 & Day 16 at 24 hours post-dose, Cycle 2 & 4 Day 1 pre-dose, EOI, Day 8 pre-dose then 7 days post last infusion (a cycle is 21 days)
  Pharmacokinetics (PK) of INI-4001 in blood plasma following multiple doses
Single dose PK Parameters - Area under the concentration-time curve (AUC0-t) | Cycle 1 Day 1 & Day 15, pre-dose, EOI (within 2 minutes), then 15 & 30 minutes, 1, 2, 4 & 6 hours post-dose, Day 2 & Day 16 at 24 hours post-dose, Cycle 2 & 4 Day 1 pre-dose, EOI, Day 8 pre-dose then 7 days post last infusion (a cycle is 21 days)
  Pharmacokinetics (PK) of INI-4001 in blood plasma following a single dose
Multiple dose PK Parameters - Area under the concentration-time curve (AUC0-t) | Cycle 1 Day 1 & Day 15, pre-dose, EOI (within 2 minutes), then 15 & 30 minutes, 1, 2, 4 & 6 hours post-dose, Day 2 & Day 16 at 24 hours post-dose, Cycle 2 & 4 Day 1 pre-dose, EOI, Day 8 pre-dose then 7 days post last infusion (a cycle is 21 days)
  Pharmacokinetics (PK) of INI-4001 in blood plasma following multiple doses
Single dose PK Parameters - Half-life (t1/2) | Cycle 1 Day 1 & Day 15, pre-dose, EOI (within 2 minutes), then 15 & 30 minutes, 1, 2, 4 & 6 hours post-dose, Day 2 & Day 16 at 24 hours post-dose, Cycle 2 & 4 Day 1 pre-dose, EOI, Day 8 pre-dose then 7 days post last infusion (a cycle is 21 days)
  Pharmacokinetics (PK) of INI-4001 in blood plasma following a single dose
Multiple dose PK Parameters - Half-life (t1/2) | Cycle 1 Day 1 & Day 15, pre-dose, EOI (within 2 minutes), then 15 & 30 minutes, 1, 2, 4 & 6 hours post-dose, Day 2 & Day 16 at 24 hours post-dose, Cycle 2 & 4 Day 1 pre-dose, EOI, Day 8 pre-dose then 7 days post last infusion (a cycle is 21 days)
  Pharmacokinetics (PK) of INI-4001 in blood plasma following multiple doses
Single dose PK Parameters - Clearance (Cl) | Cycle 1 Day 1 & Day 15, pre-dose, EOI (within 2 minutes), then 15 & 30 minutes, 1, 2, 4 & 6 hours post-dose, Day 2 & Day 16 at 24 hours post-dose, Cycle 2 & 4 Day 1 pre-dose, EOI, Day 8 pre-dose then 7 days post last infusion (a cycle is 21 days)
  Pharmacokinetics (PK) of INI-4001 in blood plasma following a single dose
Multiple dose PK Parameters - Clearance (Cl) | Cycle 1 Day 1 & Day 15, pre-dose, EOI (within 2 minutes), then 15 & 30 minutes, 1, 2, 4 & 6 hours post-dose, Day 2 & Day 16 at 24 hours post-dose, Cycle 2 & 4 Day 1 pre-dose, EOI, Day 8 pre-dose then 7 days post last infusion (a cycle is 21 days)
  Pharmacokinetics (PK) of INI-4001 in blood plasma following multiple doses
Single dose PK Parameters - Volume of distribution (Vz) | Cycle 1 Day 1 & Day 15, pre-dose, EOI (within 2 minutes), then 15 & 30 minutes, 1, 2, 4 & 6 hours post-dose, Day 2 & Day 16 at 24 hours post-dose, Cycle 2 & 4 Day 1 pre-dose, EOI, Day 8 pre-dose then 7 days post last infusion (a cycle is 21 days)
  Pharmacokinetics (PK) of INI-4001 in blood plasma following a single dose
Multiple dose PK Parameters - Volume of distribution (Vz) | Cycle 1 Day 1 & Day 15, pre-dose, EOI (within 2 minutes), then 15 & 30 minutes, 1, 2, 4 & 6 hours post-dose, Day 2 & Day 16 at 24 hours post-dose, Cycle 2 & 4 Day 1 pre-dose, EOI, Day 8 pre-dose then 7 days post last infusion (a cycle is 21 days)
  Pharmacokinetics (PK) of INI-4001 in blood plasma following multiple doses

CONTACTS AND LOCATIONS:
Overall Officials: Jon L Ruckle, Study Director — Inimmune Corp
Locations (3):
- Australia (3):
  - The Border Cancer Hospital, Albury, New South Wales
  - Southern Oncology Clinical Research Unit, Bedford Park, South Australia
  - Cabrini Hospital, Malvern, Victoria

IPD SHARING:
Plan to Share IPD: No